CLINICAL TRIAL: NCT06681701
Title: Effectiveness of Combined Manual Therapy and Pulmonary Exercises on Ventilatory Function in Patients with Restrictive Lung Diseases: a Randomized Control Trial
Brief Title: Effectiveness of Combined Manual Therapy and Pulmonary Exercises on Ventilatory Function in Patients with Restrictive Lung Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ibrahim Abuzaid, Director, Head of Department of Physiotherapy for Cardiovascular/Respiratory and Geriatrics, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Restrictive lung diseases
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Study the Effectiveness of Combined Manual Therapy and Pulmonary Exercises on Ventilatory Function in Patients with Restrictive Lung Diseases

STUDY DESIGN:
Intervention Model Description: Group B (experimental) received conventional physiotherapy and manual therapy (chest mobilization and myofascial release techniques). Treatments were performed three times weekly for 8 weeks.
  Chest mobilization (Grade III joint oscillations are administered in three bouts of thirty oscillations per second each repeated 3-5 times) was applied through the following techniques:
  Rib mobilization from sitting:
  Rib mobilization from supine:
  Central Posterior-Anterior (PA) mobilization of thoracic facet joints:
  Unilateral Posterior-Anterior mobilization of costo-vertebral joints:
  Myofascial release techniques (MRT) applied through the following (MRT was applied for 3min for each release.).
  Diaphragmatic myofascial release (DMR):
  Pectoralis minor myofascial release:
  Pectoralis major and pectoral fascia myofascial release:
  Sternocleidomastoid myofascial release:
  Scalene muscle and neck fascia myofascial release:
  Mobilize one side of the chest:
Who Masked: Participant
Masking Description: Group A (control) received conventional physiotherapy in the form of deep breathing exercises (diaphragmatic, apical, lower costal), Intensive spirometery (improve deep inspiration) and active range of motion (AROM) of both upper extremities.
  Diaphragmatic breathing exercise: S
  Segmental breathing exercises (apical, upper lateral, lower lateral and posterior basal), according to site of consolidation:
  Active Cycle Breathing Technique (ACBT):
  Intensive spirometry: It encourages patients to take deep breaths, which helps to expand the lungs and prevent complications such as pneumonia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group B (experimental) (Experimental): Group B (experimental) received conventional physiotherapy and manual therapy
  Rib mobilization from sitting:
  Rib mobilization from supine:
  Unilateral Posterior-Anterior mobilization of costo-vertebral joints:
  Myofascial release techniques (MRT)
  Diaphragmatic myofascial release (DMR):
  Pectoralis minor myofascial release:
  Pectoralis major and pectoral fascia myofascial release:
  Sternocleidomastoid myofascial release:
  Scalene muscle and neck fascia myofascial release:
  Mobilize one side of the chest:
  Interventions: Procedure: Combined Manual Therapy and Pulmonary Exercises
- Group A (control) (Active Comparator): Group A (control) received conventional physiotherapy
  Diaphragmatic breathing exercise:
  Segmental breathing exercises (apical, upper lateral, lower lateral and posterior basal), according to site of consolidation:
  Active Cycle Breathing Technique (ACBT):
  Intensive spirometry: It encourages patients to take deep breaths, which helps to expand the lungs and prevent complications such as pneumonia.
  Interventions: Procedure: Combined Manual Therapy and Pulmonary Exercises

INTERVENTIONS:
Procedure: Combined Manual Therapy and Pulmonary Exercises — Diaphragmatic breathing exercise:
  Segmental breathing exercises (apical, upper lateral, lower lateral and posterior basal), according to site of consolidation:
  Active Cycle Breathing Technique (ACBT):
  Intensive spirometry: It encourages patients to take deep breaths, which helps to expand the lungs and prevent complications such as pneumonia.
  Rib mobilization from sitting:
  Rib mobilization from supine:
  Central Posterior-Anterior (PA) mobilization of thoracic facet joints:
  Unilateral Posterior-Anterior mobilization of costo-vertebral joints:
  Diaphragmatic myofascial release (DMR):
  Pectoralis minor myofascial release:
  Pectoralis major and pectoral fascia myofascial release:
  Sternocleidomastoid myofascial release:
  Scalene muscle and neck fascia myofascial release:
  Mobilize one side of the chest:

SUMMARY:
This research investigates the effect of selective manual therapy techniques on chest expansion, pulmonary function (FVC, FEV1, and FEV1/FVC ratio), and functional capacity, in restrictive lung disease patients. The research hypothesis will be that no statistically significant difference would be found between manual therapy combined to conventional treatment and conventional treatment alone in restrictive lung disease patients.

DETAILED DESCRIPTION:
A chest physician diagnosed 72 subjects with mild to moderate restrictive lung diseases based on history, physical examination, and a ratio of FEV1/FVC above 80%. Male subjects meeting the following criteria will be included: age ranged from 50 to 60 years, BMI was 18-25 kg/m2, If a patient had a history of hiatus hernia, substantial gastro-esophageal reflux, osteoporosis, acute cardiac events within the last six weeks, congestive heart failure, acute exacerbation, exacerbation six months before, active hemoptysis, or malignant disease, they will be excluded from the study.

The subjects who consented to will be involved and met the recruitment standards randomly assigned. A computer-generated block randomization program will be used. To eliminate bias between groups, the subjects will be randomized into four-person blocks with a 1:1 allocation ratio. To ensure disguised allocation, the randomization code will be maintained in sealed, opaque envelopes consecutively numbered. A single external party will be responsible for administering the randomization

ELIGIBILITY:
Inclusion Criteria:

Restrictive lung diseases pneumonia pulmonary edema pleural effusion pneumothorax

Exclusion Criteria:

hiatus hernia substantial gastro-esophageal reflux acute cardiac events osteoporosis congestive heart failure active hemoptysis malignant disease

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function tests: Assessed by a previously calibrated portable spirometer was used (Niscomed Contec automated spirometer, 97LX89WX36mm). It is a valid test with higher reliability, as ICC = 0.912 for FVC, ICC = 0.953 for FEV1, and ICC = 0.874 for | Eight weeks
  Pulmonary function tests: Assessed by a previously calibrated portable spirometer was used (Niscomed Contec automated spirometer, 97LX89WX36mm). It is a valid test with higher reliability, as ICC = 0.912 for FVC, ICC = 0.953 for FEV1, and ICC = 0.874 for the FVC/FEV1 ratio. Subjects were advised to sit on a backrest chair, wear a nose clip, inhale deeply, hold the breath, and then exhale through a mouthpiece linked to the spirometry.2: Assessed by a previously calibrated portable spirometer was used (Niscomed Contec automated spirometer, 97LX89WX36mm). It is a valid test with higher reliability, as ICC = 0.912 for FVC, ICC = 0.953 for FEV1, and ICC = 0.874 for the FVC/FEV1 ratio. Subjects were advised to sit on a backrest chair, wear a nose clip, inhale deeply, hold the breath, and then exhale through a mouthpiece linked to the spirometry.2

SECONDARY OUTCOMES:
Assessment of Chest Expansion and Mobility | Eight weeks
  Assessment of Chest Expansion and Mobility: Assessing chest expansion and mobility is crucial for evaluating respiratory function and identifying potential chest wall pathologies. Use a non-stretchable measuring tape to assess chest expansion at three key levels: 2nd Intercostal Space (supramammary area), 4th Intercostal Space (mammary area) and Xiphoid Process (inframammary area). To measure, have the patient exhale fully to establish a baseline measurement, and then instruct them to inhale deeply. Measure the circumference at each level during full inhalation and exhalation. Compare the measurements from both sides of the chest. Normal findings should show symmetric expansion. If one side expands less than the other, it may indicate underlying issues such as lung volume loss or obstruction. Decreased expansion on one side can suggest conditions like pleural effusion, pneumothorax, or lung consolidation. Observing the mediastinum's position can also provide insights; for instance, a

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chilhate PK, Lalwani L. Manual Therapy Interventions in Patients With Chronic Obstructive Pulmonary Disease: A Comprehensive Narrative Review. Cureus. 2024 Jun 17;16(6):e62511. doi: 10.7759/cureus.62511. eCollection 2024 Jun. PMID 39022457
- [Background] Wang L, Wu X. Clinical Effects of Exercise Combined with Respiratory Training in the Rehabilitation Treatment of Patients with Chronic Obstructive Pulmonary Disease. Altern Ther Health Med. 2024 Aug;30(8):188-194. PMID 38064596